# Subject information for participation in medical research

The impact of psilocybin on pain

The impact of psilocybin on pain in fibromyalgia patients: a multicenter trial

#### Introduction

Dear Sir/Madam,

With this letter, we would like to ask you to take part in a medical study. Participation is voluntary. You have received this letter because you have been diagnosed with fibromyalgia.

You can read about the medical study in this information sheet, what it means for you, and what the pros and cons are. It is a lot of information. Can you please read the information and decide if you want to take part? If you want to take part, complete the form in **Appendix D**.

## Ask your questions

You can take your decision based on the information in this information sheet. We also suggest that you do this:

- Ask your questions to the investigator who gave you this information.
- Talk to your partner, family or friends about this study.
- Ask questions to the independent expert, Dr. Martin van Boxtel. For contact details, go to appendix A.
- Read the information on www.rijksoverheid.nl/mensenonderzoek.

## 1. General information

Maastricht University has set up this study. Below, we always call Maastricht University the 'client'. This study needs 35 subjects that completed the study in full. Participants in a medical research study are often called subjects. Both patients and people who are healthy can be subjects. The Medical Ethics Review Committee of the Academisch Ziekenhuis Maastricht (METC azM/UM) has approved this study. The research will be conducted at Maastricht University and at the Leiden University Medical Center (LUMC).

## 2. What is the purpose of the study?

In this study, we look at how safe small doses (5 and 10 mg) of psilocybin are for treating fibromyalgia. And how well it works. We compare the effect of psilocybin with the effect of a placebo. A placebo is a drug with no active ingredient, a "fake drug".

# 3. What is the background of the study?

Fibromyalgia is a long-term condition characterized by widespread pain that is often accompanied by emotional suffering (e.g., anxiety, poor mood or depression), sleep problems and disorders in memory and attention. Moreover, it is considered a condition that is difficult to treat, as most proposed treatments produce only minor improvements.

There is evidence that psychedelics (such as psilocybin), may have an analgesic effect and cause pain to be better tolerated. However, these effects have not yet been scientifically studied.

## 4. What happens during the study?

How long will the study take?

Are you taking part in the study? It will take approximately 5 weeks in total.

Step 1: are you eligible to take part?

We first want to know if you are suitable to participate. Therefore, the researcher does a number of tests.

- Before you can participate in this study, a medical screening of about 90 minutes will take place. The medical screening is based on a number of criteria regarding whether or not you can participate in the study (due to possible medical reasons). After this you will complete a questionnaire about your medical history, and a questionnaire about past and present drug and alcohol use. This will take about 30 minutes. You will then be physically examined by a physician who will ask you about your medical history. This is similar to a comprehensive sports examination, which includes taking blood (10 ml) and a urine sample. These are used for standard analyses (liver, liver, heart and kidney functions) in addition to a check for illegal drug use. In women, the urine sample is also used to test for possible pregnancy. Next, an electrocardiogram (ECG), a test that measures the electrical activity of your heartbeat, is taken.
- You will be informed if there are medical reasons why you cannot participate in this study. If you do not want to be informed of these results, you cannot participate in this study.
- Please note that it may happen that you are healthy, but you are still not suitable to participate. The researcher will tell you more about this.
- If this visit reveals that you are unable to continue participating in the study, all data and body material collected up to that point will be destroyed.

## Step 2: treatments

You will receive 3 treatments during the course of the study, one per each test day: psilocybin (5 mg), psilocybin (10 mg) and placebo. The order in which you will receive the treatment will be randomly decided.

| Possible order | Test day 1 (Visit 3) | Test day 2 (Visit 4) | Test day 3 (Visit 5) |
|---|---|---|---|
| 1 | Psilocybin – 5 mg | Psilocybin – 10 mg | Placebo |
| 2 | Psilocybin – 5 mg | Placebo | Psilocybin – 10 mg |
| 3 | Placebo | Psilocybin – 5 mg | Psilocybin – 10 mg |

Both you and the investigator will not know what treatment you received. But if this is important for your health, we can find out.

### Step 3: visit and measurements

If the screening shows that you are eligible to continue participating in the study, we will invite you to the remaining visits:

- 2nd Visit Training session (1h). During the second visit you will carry out these activities:
  - The various computer tests that you will need to perform during the examination will be practiced with you.
  - Study procedures will be explained and demonstrated to you.
- 3rd-5th Visit Test days (7h each). Between each test day there are at least 5 days when you will not receive anything, to make sure that the effects of the previous treatment are gone before you participate in the next test day. During test days you will carry out these activities:
  - Administration of psilocybin or placebo.
  - Drug test.
  - Alcohol test.
  - Pregnancy test (for women).
  - 8 Blood draws. To perform them, an IV will be inserted to avoid multiple piercing of the skin.
  - Measurement of heart rate and blood pressure
  - Several computer tasks.
  - Completion of several questionnaires. Tests that measure sensitivity to pain. Listening
    to a recorded hypnotic induction designed to produce analgesia. During the induction,
    a voice will guide you to direct your attention towards images, bodily sensations, and
    ideas.
- 6th Visit Post-study visit (1h). This follow-up measurement takes place approximately 1 week after the last test day. You fill out a number of questionnaires on the computer at home. You do not have to come to the research location for this.

See appendix C for an overview of all 5 weeks of the study and treatment day schedule.

# 5. What agreements do we make with you?

We want the study to go well. That is why we want to make the following agreements with you:

- You go to every appointment.
- You are not also participating in another medical science study during this study.
- You are not allowed to drive a traffic vehicle or to operate machines within 24 h after substance administration. This also means that you are not allowed to drive home after testing.
- From one week before the medical examination until after the follow-up visit you may not use any drugs. When drug use is detected by urine screening you will be excluded from participation.
- You must be willing to refrain from caffeine (coffee, black or green tea, or energy drink) from the evening before each visit as well as during the study day.
- You are asked to not make any substantial changes in your diet.
- You should contact the investigator in these situations:
  - You want to start taking other medication. Also, if these are homoeopathic remedies, natural remedies, vitamins or over-the-counter medicines.
  - o You are hospitalised or get treatment in a hospital.
  - o You suddenly have problems with your health.
  - You no longer want to take part in the study.
  - o Your telephone number, address or email address changes.

Is it OK for you or your partner to get pregnant during the study?

Women who are pregnant or breastfeeding cannot take part in this study. Women should also not get pregnant during the study. Are you male and do you have a female partner? Then you need to make sure that she cannot become pregnant with your child.

In fact, this research may have implications for an unborn child. It is not known what consequences. The investigator will tell you how best to prevent pregnancy. Talk to your partner about this.

#### Pregnant after all?

Will you become pregnant during the study? Please inform the medical examiner immediately. In consultation with the researcher, you should then stop this study as soon as possible.

## 6. What side effects, adverse effects or discomforts could you experience?

The substance to be investigated may cause adverse effects. You will be given psilocybin in small doses with possible mind-altering properties. Psilocybin may influence your feelings (excitement, joy but also fear and panic) and perception. Psilocybin can cause a distortion of time and space and alter the perception of your own body.

The following side effects are common:

#### Increased heart rate

#### Measurements

Blood draws may cause pain or bruising, which normally heals within 2 to 3 days. In rare cases, blood clots may form or veins may become inflamed.

In total, we will draw about 190 ml of blood from you. This amount should not cause any problems in adults. In comparison, at the blood bank, 500 mL of blood is collected at one time.

Finally, filling questionnaires can be tiring.

# 7. What are the pros and cons if you take part in the study?

Taking part in the study can have pros and cons. We will list them below. Think about this carefully and talk to other people about it.

If you take part to the study, you may experience a pleasant alteration of your state of mind and psilocybin may reduce pain intensity although it is not certain. But your participation will help in the search for a possible treatment for fibromyalgia in adults.

Taking part in the study can have these cons:

- You may experience the adverse effects of psilocybin, as described in section 6.
- There may be some discomfort from the measurements during the study. For example: taking a blood sample can be a little painful or you could get a bruise as a result and the pain task will require you to submerge your hand in very cold water.
- Taking part in the study will cost you extra time.
- You have to comply with the study agreements.

You do not wish to participate in the study?

It is up to you to decide if you wish to participate in the study. Participation is voluntary.

## 8. When does the study end?

The researcher will let you know if there is any new information about the study that is important to you. The researcher will then ask you if you want to continue to take part.

In these situations, the study will stop for you:

- All checks according to the schedule are finished.
- The end of the whole study has been reached.
- You have become pregnant.
- You want to stop participating in the study yourself. You can stop at any time. Report this to
  the investigator immediately. You do not have to explain why you want to stop. The
  investigator will still contact you for a follow-up check.
- The investigator thinks it is better for you to stop. The investigator will still contact you for a follow-up check.

- One of the following authorities decides that the study should stop:
  - Maastricht University,
  - o the government, or
  - the Medical Ethics Review Committee assessing the study

What happens if you stop participating in the study?

The investigators use the data and blood samples that have been collected up to the moment that you decide to stop participating in the study. If you wish, we will destroy the collected body material. Please let the investigator know.

The entire study ends when all the participants have finished.

# 9. What happens after the study has ended?

Will you get the results of the study?

About one year after the study has ended, the investigator will inform you about the most important results of the study. The investigator may also tell you in what order you received the treatments. Do you prefer not to know? Please tell the investigator. You can indicate your preference on the Informed Consent form, in **appendix D**.

# 10. What will be done with your data and body material?

Are you taking part in the study? Then you also give your consent to collect, use and store your data and body material. The body material may be used by the sponsor and laboratories that assist the sponsor in analysing the body material.

What data do we store?

We store these data:

- your name
- your gender
- your address
- your date of birth
- information about your health
- (medical) information that we collect during the study

What body material do we store?

We collect, use and store blood samples.

Why do we collect, use and store your data and body material?

We collect, use and store your data and your body material to answer the questions of this study and to be able to publish the results.

How do we protect your privacy?

To protect your privacy, we give a code to your data and your body material. We only put this code on your data and body material. We keep the key to the code in a safe place at the university. When we process your data and body material, we always use only that code. Even in reports and publications about the study, nobody will be able to see that it was about you.

## Who can see your data?

Some people can see your name and other personal information without a code. This could include data specifically collected for this study, but also data from your medical file. These are people checking whether the investigators are carrying out the study properly and reliably. These persons can access your data:

- A controller working for the sponsor.
- National and international supervisory authorities. For example, the Inspectorate for Healthcare and Youth.

These people will keep your information confidential. We ask you to give permission for this access. The Health and Youth Inspectorate can access your personal information without your permission.

For how long do we store your data and body material?

We will store your data at Maastricht University for 25 years. The body material will be destroyed once analyses are complete.

## Can we use your data for other research?

Your data may also be important after this study for other scientific research on the analgesic effects of psilocybin. For this purpose, your data will be stored at Maastricht University for 25 years. Please indicate in the consent form whether you agree with this. Do you not want to give your consent? Then you can still take part in this study.

### What happens if there are coincidental findings?

It is possible that during the study we discover something that is not directly relevant to the study but is important for your health or for the health of your family members. The medical examiner will then contact your general practitioner (GP). You will then discuss with your GP or specialist what needs to be done. By submitting this form, you grant permission for your GP or specialist to be informed.

## Can you take back your consent for the use of your data?

You can take back your consent for the use of your data at any time. Please tell the investigator if you wish to do so. This applies both to the use in this study and to the use in other medical research. But please note: if you take back your consent, and the investigators have already collected data for research, they are still allowed to use this information. The investigators will destroy your body material after you take back your consent. But if assessments with your body material have been carried out, the investigator can continue to use the results.

Do you want to know more about your privacy?

- Do you want to know more about your rights when processing personal data? Visit www.autoriteitpersoonsgegevens.nl.
- Do you have questions about your rights? Or do you have a complaint about the processing of your personal data? Please contact who is responsible for processing your personal data. For the present study, this is Maastricht University. See appendix A for contact details, and website.
- If you have any complaints about the processing of your personal data, we recommend that
  you first discuss them with the research team. You can also contact the Data Protection
  Officer of Maastricht University. Or you can submit a complaint to the Dutch Data Protection
  Authority.

Where can you find more information about the study?

You can find more information about the study on the following website: <a href="www.trialregister.nl">www.trialregister.nl</a> After the study, the website may show a summary of the results of this study. You can find the study by searching for number NL78008.068.21.

# 11. Will you receive compensation if you participate in the study?

You will receive € 225 for participation in the whole study. This is based on € 10/hour, plus € 15 bonus if you participate in all conditions. In case of premature termination of the study, compensation will be based on the number of hours. In addition, tickets for using public transport to come to the test site and to return home will be reimbursed. The compensation for taking part in this study may need to be declared to the Tax and Customs Administration as 'income from other resources'. If necessary ask the Tax services.

# 12. Are you insured during the study?

Insurance has been taken out for everyone who takes part in this study. The insurance pays for damage caused by the study. But not for all damage. You can find more information about this insurance and any exceptions in **appendix B**. It also says who you can report damage to.

## 13. We will inform your doctor.

The investigator will send your doctor an email to let them know that you are taking part in the study. This is for your own safety.

## 14. Do you have any questions?

You can ask questions about the study of the research team. Would you like to get advice from someone who is independent from the study? Then contact Dr. Martin van Boxtel. He knows a lot about the study, but is not a part of this study.

Do you have a complaint? Discuss it with the investigator or the doctor who is treating you. If you prefer not to do so, please contact the Complaints Commission. **Appendix A** provides the contact details.

# 15. How do you give consent for the study?

You can first think carefully about this study. We ask you to take at least one week to consider whether you wish to participate. Then you can tell the investigator if you understood the information, whether you have any question regarding the study and if you want to take part or not. If you want to take part, you will be given an appointment where you will be able to fill in the consent form (**appendix D**) and sign it at the presence of the investigator. You and the investigator will both get a signed version of this consent form.

Thank you for your attention.

# Appendices to this information

- A. Contact details for the study at Maastricht University
- B. Information about the insurance
- C. Overview and description of study interventions
- D. Consent form

# Appendix A. Contact details for Maastricht University

Visiting address:

Maastricht University

Faculty of Psychology & Neuroscience

Department of Neuropsychology & Psychopharmacology
Universiteitssingel 40, 6229 ER Maastricht

Principal Investigator:
Prof. Dr. Johannes .G. Ramaekers
Maastricht University
Tel. +31 43 3881951
Email: j.ramaekers@maastrichtuniversity.nl

Independent Expert:
Dr. Martin van Boxtel
Maastricht University
Tel. (043) 38 81028
martin.vanboxtel@maastrichtuniversity.nl

Medical Supervisor: Cees van Leeuwen Maastricht University Tel. 06-5144 6431

Complaints Officer: Rense Hoekstra Maastricht University Tel. (043) 38 84539

Email: rense.hoekstra@maastrichtuniversity.nl

For more information about your rights: Data Protection Officer of the institution: Email: fg@maastrichtuniversity.nl

Website: https://www.maastrichtuniversity.nl/nl/over-de-um/algemene-privacyverklaring-um/ontvangers-van-persoonsgegevens

Study Coordinator and Contact Person Mauro Cavarra Maastricht University Tel. (043) 38 83517 Email: fpn-pim\_p137@maastrichtuniversity.nl

During working hours you can reach us at the university: (043) 388 3517 (Mauro Cavarra).

In an **emergency** outside working hours: 043-38 84017. Through this phone number, you can reach out to any of the researchers 24 hours a day 7 days a week.

# Appendix B. Information about the insurance

The University of Maastricht has taken out insurance for everyone who takes part in the study titled *The impact of psilocybin on pain in fibromyalgia patients: a multicenter trial.* The insurance pays for the damage you have suffered because you participated in the study. This concerns damage you suffer during the study or within 4 years after the study has ended. You must report damage to the insurer within 4 years.

Have you suffered damage as a result of the study? Please report this to this insurer or the contact person at Maastricht University. See the contact details below.

The insurer of the study is:

Name: CNA Insurance Company Europe S.A.

Address: Polarisavenue 140, 2132 JX Hoofddorp, The Netherlands

(Policy number: 10378335)

The Broker Liability of the study is:

Name: Youri (Y.C.) de Goeij, AON Commercial Risk Solutions

Address: Administratiekade 62, 3063 ED Rotterdam, The Netherlands

Email: youri.de.goeij@aon.nl

Telephone number: +31 (0)6 547 759 64

The contact person at Maastricht University is:

Name: department Treasury, Linda Lemmens

Address: Maastricht University, Postbus 616 6200 MD Maastricht, The Netherlands

Email: um-verzekeringen@maastrichtuniversity.nl

Telephone number: +31 (0)6 287 443 61

The insurance pays a maximum of at least €650,000 per person and at least €5,000,000 for the entire study (and € 7,500,000 per year for all studies by Maastricht University).

Please note that the insurance does **not** cover the following damage:

- Damage due to a risk about which we have given you information in this sheet. But this does
  not apply if the risk turned out to be greater than we previously thought. Or if the risk was very
  unlikely.
- Damage to your health that would also have happened if you had not taken part in the study.
- Damage that happens because you did not follow directions or instructions or did not follow them properly.
- Damage to the health of your children or grandchildren.
- Damage caused by a treatment method that already exists. Or by research into a treatment method that already exists.

These provisions can be found in the 'Besluit verplichte verzekering bij medisch-wetenschappelijk onderzoek met mensen 2015' ('Medical Research (Human Subjects) Compulsory Insurance Decree 2015'). This decision can be found in the Government Law Gazette (<a href="https://wetten.overheid.nl">https://wetten.overheid.nl</a>).

## Appendix C. Overview and description of study interventions

## Inclusion criteria for the study include:

- Age between 18 and 65 years
- Normal weight, body mass index (weight/height2) between 18 and 28 kg/m2
- Fulfilment of the American College of Rheumatology criteria for FM diagnosis [43]
- A minimum NRS pain score of 5 out of 10
- Proficient knowledge of the Dutch or English language
- Written Informed Consent
- Understanding the procedures and the risks associated with the study
- No regular use of psychotropic medication such as opiates, antidepressants, muscle relaxants, anticonvulsants, sleep aids, benzodiazepines. Non pharmacological regimens will be allowed along with 1 rescue therapy such as acetaminophen ≤4,000 mg/day, ibuprofen ≤1,200 mg/day, naproxen ≤660 mg/day, or ketoprofen ≤75 mg/day. Use of paracetamol (PCM) and non-steroidal anti-inflammatory drugs (NSAIDS) will be allowed.
- Willingness to refrain from taking psychoactive substances during the study.
- Willingness to drink only alcohol-free liquids and no coffee, black or green tea, or energy
  drinks after midnight of the evening before the study session, as well as during the study days
- Willingness not to drive a traffic vehicle or to operate machines within 24 h after substance administration

### **Exclusion criteria for this study include:**

- Presence of any other painful condition such as inflammatory rheumatic diseases, migraines
  or headaches and of other chronic or acute medical conditions
- Presence or history of any other psychiatric condition such as primary major depressive disorder, anxiety disorders or substance use disorder as determined by the medical questionnaire, drug questionnaire and medical examination
- Previous experience of serious side effects to psychedelic drugs (anxiety or panic attacks)
- Tobacco smoking (>20 per day)
- Excessive drinking (>20 alcoholic consumptions per week)
- Psychotic disorder in first-degree relatives
- Pregnancy or lactation
- Hypertension (diastolic > 90 mmHg; systolic > 140 mmHg)
- History of cardiac dysfunctions (arrhythmia, ischemic heart disease...)
- For women: no use of a reliable contraceptive

Below you will find tables summarising the visits and the schedule of each test day visit.

| Table 1. Visits, duration | Table 1. Visits, duration and summary of activities | | |
|---|---|---|---|
| Timepoint | Visit | Time | Content |
| Visit 1 | Consent and medical screening | ±45 min | Information about the study, consent, drug questionnaire, medical questionnaire. Medical and psychological examination. Blood samples (10ml) for laboratory analysis, pregnancy and drug tests. |
| Visit 2 | Training session | 1 hour | Memory and attention tasks,<br>questionnaires and study<br>procedures explained |
| Visit 3 | Test day 1 | 7 hours | Administration with psilocybin (5 mg or 10 mg) or placebo. Pregnancy and drug test, alcohol test, blood samples, questionnaires, tasks. |
| Visit 4 | Test day 2 | 7 hours | Administration with psilocybin (5 mg or 10 mg) or placebo. Pregnancy and drug test, alcohol test, blood samples, questionnaires, tasks. |
| Visit 5 | Test day 3 | 7 hours | Administration with psilocybin (5 mg or 10 mg) or placebo. Pregnancy and drug test, alcohol test, blood samples, questionnaires, tasks. |

| Visit 6 (online) | Post-study visit | 1 hour | Administration of post-study measures |
|---|---|---|---|

| | | 10.00 | 10.30 | 11.00 | 11.30 | 12.00 | 12.30 | 13.00 | 14.00 | 15.00 | 16.00 |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Table 1. Schedule of events for | each | session | | | | | | | | | |
| Relative Time | -1 | 0 | 0.5 | 1 | 1.5 | 2 | 2.5 | 3 | 4 | 5 | 6 |
| Substance Administration | | | | | | | | | | | |
| Psilocybin/Placebo | | X | | | | | | | | | |
| Pain | | | | | | | | | | | |
| PPT | | | | | 1 | | | | 2 | | |
| CPT | | | | | 1 | | 2* | | 3 | | |
| BPI | | | | | | | | | | | 1 |
| Psychometrics | | | | | | | | | | | |
| VAS | 0 | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 |
| POMS | 0 | | | 1 | | 2 | | 3 | | 4 | |
| CADSS, BSI | 0 | | | | | | | | | | 1 |
| 5D-ASC, EDI | | | | | | | | | | | 1 |
| Autonomic Measures | | | | | | | | | | | |
| BP, HR | -1 | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 |
| Blood samples | | | | | | | | | | | |
| Substance concentration | 0 | | 1 | 2 | 3 | 4 | | 5 | 6 | | 7 |
| BDNF | 0 | | | | | 1 | | | 2 | | 3 |
| Computer tests | | | | | | | | | | | |
| ART | | | | | | | | | | 1 | |
| MET | | | | 1 | | | | | | | |
| Story Writing | | | | | | 1 | | | | | |
| AUT | | | | | | | 1 | | | | |
| AMT | | | | | | | | | | 1 | |
| DSST, PVT | | | | | 1 | | | | 2 | | |

Visual Analogue Scale (VAS), Profile of Mood States (POMS), Clinical Administered Dissociative States Scale (CADSS), Brief Symtpoms Inventory (BSI), Altered States of Consciousness (5D-ASC), Ego Dissolution Inventory (EDI), Blood pressure (BP), Heart rate (HR), Multifaceted Empathy Test (MET), Alternate Use Test (AUT), Digit Symbol Substitution Test (DSST), Psychomotor Vigilance Task (PVT), Pressure Pain Threshold (PPT), Cold Pressor Task (CPT), Brief Pain Inventory (BPI), Autobiographical Recollection Test (ART).

Description of the various tests and questionnaires, which will be administered during the examination:

• **Psilocybin/placebo**: the administration of psilocybin or placebo will occur on test days around 10.00.

<sup>\*</sup> CPT plus suggestion

- **PPT** Pain Pressure Threshold: we will apply an algometer (a tool to measure pressure-related pain sensitivity). The algometer has a small circular head that will be pressed against your hand. The experimenter will increase pressure until you will feel pain and then stop. That pressure value will be recorded and used for analysis.
- CPT Cold Pressor Test: you will be asked to submerge your hand in cold water and
  to keep it there for as long as you can. You will be asked to report when you will start
  to feel pain and, once the test is over, to report on a scale from 0 to 10 how painful,
  unpleasant and stressful the experience was. In conjunction with the second CPT
  administration, you will be asked to listen to a recorded hypnotic induction containing
  suggestions designed to promote analgesia.
- **BPI** Brief Pain Inventory: a questionnaire that assesses pain severity and interference in your daily life.
- **VAS** Visual Analogue Scale: you will be asked to rate how much you do feel under the effect of psilocybin/placebo on a scale ranging from "not at all" to "extremely".
- POMS Profile of Mood States: a questionnaire that assesses your mood and emotional state.
- **CADSS** Clinician Administered Dissociative States Scale: a questionnaire that assesses dissociative symptoms (e.g., depersonalisation, derealisation).
- BSI Brief Symptom Inventory: a questionnaire that assesses the presence of depressive, anxious and somatization symptoms.
- **5D-ASC** 5 Dimension Altered States of consciousness: a questionnaire that assesses the effects of psychedelic substances.
- EDI Ego Dissolution Inventory: a questionnaire assessing ego dissolution experiences. These experiences are sometimes reported as a consequence of psychedelic intake and are described as a feeling of being one with the universe and of losing one's boundaries.
- **BP & HR** Blood Pressure and Heart Rate: through the use of an electronic device, we will regularly monitor these two parameters.
- **Substance concentration**: we will periodically draw samples through a cannula that will be placed at the beginning of the study day. These samples will be used to assess substance concentration at different times after administration.
- **BDNF** Brain Derived Neurotrophic Factor: BDNF is a substance that can be detected in the bloodstream. Higher concentrations of it are associated with improved neuroplasticity, which is the capacity of the brain to form new connections.
- MET Multifaceted Empathy Test: a computerised test that assesses empathy,
  defined as the ability to infer the mental states of others. You will be shown images of
  people in emotionally charged situations and be asked to identify their mental state
  and to report how much you feel for them and how much you are aroused by the
  scene.
- **Story writing**: a task designed to assess creativity. You will be asked to write a story from three words that will be assigned to you during the study day.

- AUT Alternate Use Test: a task designed to assess creativity. You will be asked to
  list as many possible uses you can come up with of 3 everyday objects in a fixed
  timespan.
- DSST Digit Symbol Substitution Test: a computerised test designed to assess
  cognitive function. You will be shown a legend that pairs each symbol from a
  determined list with a number from 1 to 9. Subsequently, you will be presented an
  array of symbols and you will be asked to write the corresponding number under each
  symbol as fast as you can.
- PVT Psychomotor Vigilance Task: a computerised task designed to measure vigilance. You will be asked to press a button as quickly as possible when a prompt will appear on the screen.
- AMT Autobiographical Memory Test: Based on cue words that will be provided, you will be asked to recall memories of events in your past.
- ART Autobiographical Recollection Test: you will be asked to respond to a set of questions about how you remember personal events.

# Appendix D. Informed consent form – subject

Belonging to

The impact of psilocybin on pain

- I have read the information sheet. I was able to ask questions. My questions have been answered well enough. I had enough time to decide if I wanted to take part.
- I know that participation is voluntary. I also know that at any time I can decide not to participate in the study. Or to stop. I do not have to say why I want to stop.
- I give the investigator consent to inform my doctor that I am taking part in this study.
- I give consent to give my doctor or specialist information about accidental discoveries made during the study that are important for my health.
- I give consent to collect and use my data and blood samples. The investigators only do this to answer the questions of this study.
- I know that some people will be able to see all of my data to review the study. These people
  are mentioned in this information sheet. I give consent to let them see my data for this review.
- I know that I cannot get pregnant/cannot get my partner pregnant during the study.
- The investigator discussed with me how I can best prevent becoming pregnant/my partner from becoming pregnant.
- I am aware that my anonymized study data will be shared with Usona Institute. I know that this data is not in any way traceable back to my personal data.
- Please tick yes or no in the table below.

| I give consent to store my data to use for other research, as stated in the | Yes | No |
|---|---|---|
| information sheet. | | |
| I give consent to let me know after the study which treatment I received/in which | Yes | No |
| group I was. | | |
| I give consent to ask me after this study if I want to participate in a follow-up study. | Yes | No |

| - I want to take part in this study. | | |
|--------------------------------------|------|-----|
| My name is (subject):Signature: | Date | :// |

I declare that I have fully informed this subject about the study mentioned.

If any information becomes known during the study that could influence the subject's consent, I will let this subject know in good time.

| Investigator name (or their representative): | |
|----------------------------------------------|---------|
| Signature: | Date:// |

The study subject will receive a complete information sheet, together with a signed version of the consent form.